CLINICAL TRIAL: NCT05646485
Title: Optimal Screening Strategy for Bladder Cancer in at Risk Patients
Brief Title: Bladder Cancer Screening Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Wilson Charitable Foundation Trust (Unknown); Pacific Edge Limited (Industry)
Responsible Party: Principal Investigator, yair lotan, Professor-Urology, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STU-2022-1042
Record Dates: First submitted 2022-12-01; First posted 2022-12-12 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Bladder Cancer; Urothelial Carcinoma; Hematuria; Smoking Cessation
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Hematuria; Smoking Cessation | interventions — Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BCa Early Screening Group (Experimental): All participants undergo Urinalysis testing every 6 months for 2 years. Based on the RBC count, each participant will go through each of the screening procedures : [cystoscopy + Upper tract imaging] or [urine marker cancer testing with Cxbladder triage + Upper tract imaging] or [Repeat urinalysis]
  Patients with suspicious findings on cystoscopy or imaging will get treatment as per standard of care.
  Their outcomes will be compared to a historical control (bladder cancer detected by standard of care using SEER registries).
  Interventions: Diagnostic Test: Urinalysis
- Historical Control Group (No Intervention): This will include historical control (bladder cancer detected in patients by standard of care) using SEER registries).

INTERVENTIONS:
Diagnostic Test: Urinalysis — Urine analysis (every 6 months for 2 years); Patients with <3 red blood cells (RBCs) per high-powered field (HPF) will repeat screening at 6-month intervals for an average of 2 years.
  If RBCs are 3-25 RBSc/HPF- subjects will undergo- [cystoscopy + Upper tract imaging] or [urine marker cancer testing with Cxbladder triage + Upper tract imaging].
  If >25 RBCs, subjects will get - [cystoscopy + Upper tract imaging].
  Arms: BCa Early Screening Group

SUMMARY:
There is currently no accepted screening strategy for patients at high risk of developing bladder cancer. This study will ask patients to complete a urine test every 6 months for 2 years to help assess if routine screening helps finding bladder cancer at an earlier stage.

DETAILED DESCRIPTION:
Bladder cancer is the 4th most common cancer in men and 6th most common cancer overall with over 80,000 new cases in the US per year. The most common causes of bladder cancer are smoking and it is usually found in patients over the age of 50. By the time it is diagnosed, the disease is often advanced since there are few warning signs other than seeing blood in the urine.

Screening is currently accepted practice for colon, cervical, and breast cancer. However, there is not an accepted screening methodology for bladder cancer. Bladder cancer is currently detected in 2-5% of patients who have microhematuria on routine urinalysis, a cheap, non-invasive test obtained by many primary care physicians. Bladder cancer diagnosed by microscopic blood on urinalysis is often lower stage than patients diagnosed with visible blood. Urine testing, therefore, offers a simple screening mechanism that can be tailored to patients at higher risk for bladder cancer based on age, tobacco exposure and other risk factors. In conjunction with routine traditional urinalysis testing, there are advances in urine molecular markers which utilize protein and genetic alterations resulting in a higher sensitivity and specificity for the detection of bladder cancer. Markers have not been evaluated for screening in high-risk populations, and there is a gap in knowledge of the most accurate screening method.

Early detection of bladder cancer has the potential to identify disease at an earlier stage resulting in a lower burden of treatment, improved quality of life, and improved survival.

This study will prospectively screen patients at high risk for the development of bladder cancer at bi-annual intervals with a commonly available urinalysis test that assess for microhematuria and urine based molecular markers.

This is a single arm study. The outcomes from the experimental arm will be compared to a historical control (bladder cancer detected by standard of care using SEER registries).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50
* Smoking: ≥15 pack-year smoking history
* Occupation:≥ 15 years of occupational exposures including: textile worker, painter, dry cleaners

Exclusion Criteria:

* Prior history of bladder, kidney, or prostate cancer
* Prior evaluation of micro or gross hematuria within the last 2 years
* Do not provide informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Bladder cancer (BCa) | 5 years
  Incidence of Bladder cancer is measured by the number of participants who were detected with BCa.

SECONDARY OUTCOMES:
Smoking cessation | 3 years
  Smoking cessation is measured by number of participants who were referred to smoking cessation treatment
Screening interval | approx. every 6 months for up to 2 years
  Screening interval is assessed by calculating the average screening interval from baseline until the timepoint when RBCs >3 are detected for each participant
Screening interval | approx. every 12 months for up to 2 years
  Screening interval is assessed by calculating the average screening interval from baseline until the timepoint when RBCs >3 are detected for each participant
Number of participants with positive/ negative markers and findings on cystoscopy | 2 years
  Performance of urinalysis and molecular markers is assessed by the count of participants with positive/ negative markers and findings on cystoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lotan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No